CLINICAL TRIAL: NCT00302042
Title: Translating the DPP Into the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ronald Ackermann, ctor, Institute for Public Health and Medicine, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DK70702 (completed); R34DK070702 (NIH)
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2014-08

CONDITIONS: Prediabetic State; Overweight; Obesity
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity | interventions — Residence Characteristics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Brief Counseling Plus Group Lifestyle (Experimental): Brief counseling plus group diabetes prevention in community
  Interventions: Behavioral: Brief counseling plus group diabetes prevention in community
- 2: Brief Counseling Alone (Active Comparator): Brief Counseling for pre-diabetes alone
  Interventions: Behavioral: Brief Counseling for pre-diabetes alone

INTERVENTIONS:
Behavioral: Brief counseling plus group diabetes prevention in community — Brief counseling at measurement visits: education about diabetes and the importance of medical follow-up for determining the most appropriate strategies to decrease this risk, Group diabetes prevention in community: 16 weekly group lifestyle behavior change visits followed by monthly group lifestyle behavior change visits.
  Arms: 1: Brief Counseling Plus Group Lifestyle
Behavioral: Brief Counseling for pre-diabetes alone — Brief counseling at measurement visits: education about diabetes and the importance of medical follow-up for determining the most appropriate strategies to decrease this risk.
  Arms: 2: Brief Counseling Alone

SUMMARY:
The Diabetes Prevention Program (DPP) demonstrated that an intensive lifestyle intervention resulting in modest weight loss and increased physical activity can delay or prevent the development of type 2 diabetes in those at increased risk for the disease. The lifestyle program used, however, was not designed for delivery on a public health scale. Successful community translation of the DPP's findings will require close collaboration with an established community organization committed to improving community health and experienced in implementing sustainable health and wellness programs. With exceptional reach into diverse U.S. communities, the Young Mens Christian Association (YMCA) may be an ideal community partner. We have been collaborating with the YMCA organization for over a year to design a robust recruitment and implementation model that is sensitive to the unique needs and resources of a community organization. We now propose to evaluate if a group-based adaptation of the DPP lifestyle intervention can be successfully implemented by YMCA staff, in YMCA facilities. We have designed this study to develop preliminary data about the reach, effectiveness, and consistent implementation of the DPP lifestyle intervention in this context. This pilot study has two primary aims: 1) to demonstrate the extent to which YMCA staff trained by DPP study personnel can administer a group-based adaptation of the DPP lifestyle intervention in a fashion consistent with DPP intervention protocols, and 2) to evaluate if the intervention program delivered by the YMCA results in changes in body mass, physical activity, and dietary intake that are consistent with a level found to be associated with diabetes risk reduction during the DPP trial. We will also collect valuable data about the feasibility and reach of a selective, community-based marketing and screening approach for recruiting program participants. In combination, these data will enable us to design and conduct a larger, future 3-year trial focusing on the effectiveness and sustainability of community DPP translation in multiple YMCA settings.

ELIGIBILITY:
Inclusion Criteria:

i. 18 years of age or older ii. Body-mass index of >= 24 kg/m2 iii. ADA diabetes risk assessment score >= 10 (see below) iv. Casual capillary blood glucose >= 110 mg/dl

Exclusion Criteria:

i. Exclusions for diseases likely to limit life span and/or increase risk of interventions:

A. Cancer requiring treatment in the past 5 years

B. Cardiovascular disease:

1. A "Yes" response to any item on the modified Physical Activity Readiness Questionnaire (see Appendix 2)
2. Uncontrolled hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >105 mmHg
3. Heart attack, stroke, or transient ischemic attack in the past 6 months, C. Lung disease: Chronic obstructive airways disease or asthma requiring home oxygen

ii. Exclusions related to metabolism: A. Diabetes at baseline evaluation B. Casual capillary blood glucose >= 200 mg/dl C. History of anti-diabetic medication use (oral agents or insulin) except during gestational diabetes

D. Pregnant female E. Self-report of disease associated with disordered glucose metabolism: Cushing's syndrome; acromegaly; pheochromocytoma; chronic pancreatitis

iii. Exclusion for conditions or behaviors likely to affect the conduct of the study:

A. Unable or unwilling to provide informed consent B. Unable to communicate with the pertinent clinic staff C. Unable to read written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2005-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald T Ackermann, MD, MPH, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Diabetes Prevention and Control Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: 1: Brief Counseling Plus Group Lifestyle: Brief counseling for pre-diabetes plus access to a group-based diabetes prevention lifestyle intervention in the community
- Active Comparator: 2: Brief Counseling Alone: Brief Counseling for pre-diabetes alone without access to group lifestyle
Period: Overall Study
Arm/Group | Experimental: 1: Brief Counseling Plus Group Lifestyle | Active Comparator: 2: Brief Counseling Alone
Started | 46 | 46
Completed | 39 | 38
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: 1: Brief Counseling Plus Group Lifestyle | Active Comparator: 2: Brief Counseling Alone | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 43 | 88
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (9.7) | 60.1 (10.5) | 58.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 23 | 18 | 41
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: 6 months minus baseline
Time Frame: Baseline, 6 months
Measure: Mean (95% Confidence Interval); unit: percentage of change in weight
Arm/Group | Experimental: 1: Brief Counseling Plus Group Lifestyle | Active Comparator: 2: Brief Counseling Alone
Number analyzed (Participants) | 39 | 38
percentage of change in weight | -6.0 [-7.3 to -4.7] | -2.0 [-3.3 to -0.6]

2. Secondary Outcome: Physical Activity Level
Time Frame: Baseline, 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Rate of Community Program Participation
Time Frame: Baseline, 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Dietary Composition
Time Frame: Baseline, 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not specifically elicited from participants in this minimal risk small pilot trial. However, none were spontaneously reported by participants.
Arm/Group | Experimental: 1: Brief Counseling Plus Group Lifestyle | Active Comparator: 2: Brief Counseling Alone
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No